CLINICAL TRIAL: NCT06507995
Title: The Effectiveness of Thoracal Epidural Steroid and Local Anesthetic Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Dostalı Alıyev, Principal Investigator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: i7-487-21
Record Dates: First submitted 2024-06-26; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Chronic Postoperative Pain; Chest Pain; Back Pain
Keywords: Chronic thoracic pain; chest wall pain; thoracic interlaminar epidural injections
MeSH Terms: conditions — Pain, Postoperative; Chest Pain; Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local Group (Other): Group I received thoracic interlaminar epidural injections of 6 mL of 2% preservative-free prilocaine.
  Interventions: Drug: thoracic interlaminar epidural injection
- Local+steroid Group (Other): Group II received injections of 4 mL of 2% preservative-free prilocaine combined with 2 mL or 8 mg of dexamethasone, totaling 6 mL
  Interventions: Drug: thoracic interlaminar epidural injection

INTERVENTIONS:
Drug: thoracic interlaminar epidural injection — . Injections were administered under sedation and sterile conditions, with all patients positioned prone and monitored. A single physician performed all injections using an 18 gauge Tuohy needle, employing the loss of resistance technique and confirming the epidural space placement with 5 mL of nonionic contrast.

SUMMARY:
The primary objective was to evaluate the effectiveness of thoracic interlaminar epidural injections in alleviating pain and enhancing function in patients suffering from chronic mid and/or upper back pain.

Materials and Methods One hundred patients were randomly divided into two groups, each consisting of 50 patients. Group I received only a local anesthetic, while Group II received a combination of local anesthetic and steroids. The random assignment to either Group I or Group II was determined using a simple computer-generated sequence.

Outcomes were evaluated using the Numeric Rating Scale (NRS) and the revised Oswestry Disability Index (rODI). Patients who showed significant improvement for more than four weeks after the first two procedures were deemed successful. Those who did not were classified as failed participants. Significant improvement was defined as a reduction of more than 50% in both NRS and rODI scores, with assessments conducted at baseline and at 3, 6, and 12 months post-treatment.

The center where the study was conducted: Ankara University, Faculty of Medicine, Department of Anesthesiology and Reanimation, Division of Algology, Ankara, Turkey

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* > 6 months pain duration
* Failed conservative management (including medication, physical therapy, and exercise programs)
* Facet joint pain ruled out (confirmed through diagnostic blocks)

Exclusion Criteria:

* < 18 years old
* Having a psychological illness
* Allergies to local anesthetics or steroids
* Thoracic facet joint pain
* Significant disc herniation
* Infection ( which were ruled out by pre-procedure blood tests and C-reactive protein levels)

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
The effect of thoracic epidural injection on upper back pain | 1 year
  Change in Visual Analog Score after the procedure. The visual analog scale (VAS) of pain intensity consists of a line, most often 100 mm long, with 2 descriptors representing extremes of pain intensity (eg, no pain and extreme pain)at each end. The findings suggested that 100-mm VASratings of 0 to 4 mmcanbeconsidered nopain; 5 to 44mm,mildpain; 45 to 74mm, moderate pain; and 75 to 100 mm, severe pain.
The effect of thoracic epidural steroid and local anesthetic injection on upper back pain | 1 year
  Change The Oswestry Disability Index (ODI) after the procedure:
  ODI is an index used by clinicians and researchers to quantify disability for low back pain and quality of life. The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible. 0% -20%: Minimal disability;21%-40%: Moderate Disability;41%-60%: Severe Disability;61%-80%: Crippling back pain;81%-100%;The patient is either bed-bound or has an exaggeration of their symptoms.

SECONDARY OUTCOMES:
The effect of thoracic epidural steroid and local anesthetic injection on upper back pain | 1 year
  Body mass index difference between groups
The effect of thoracic epidural steroid and local anesthetic injection on upper back pain | 1 year
  Difference between groups in duration of pain
The effect of thoracic epidural steroid and local anesthetic injection on upper back pain | 1 year
  Gender difference between groups

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)